CLINICAL TRIAL: NCT04884516
Title: Study to Identify if Embody's Retinol Gummy Works to Improve the Appearance of Early Signs of Aging and to Examine if it Reduces the Overall Frequency and Intensity of Adult Acne.
Brief Title: Study To Investigate If Embody's Retinol Gummies Improve The Early Signs Of Skin Aging And Overall Skin Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Embody Beauty, Inc. (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EmbodyRetinol
Record Dates: First submitted 2021-05-06; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Acne, Adult
Keywords: skin aging; adult acne
MeSH Terms: conditions — Acne, Adult; Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Other): Participants take retinol gummy once a day
  Interventions: Dietary Supplement: Retinol gummy

INTERVENTIONS:
Dietary Supplement: Retinol gummy — Participants take one retinol gummy per day

SUMMARY:
The Embody retinol study is a single-arm clinical trial on skin aging prevention and adult acne. The purpose of this study is to determine the effect of a retinol gummy in adults aged 18-45 on skin aging and overall skin health.

DETAILED DESCRIPTION:
Embody has developed a retinol gummy with the aim to improve the appearance of early signs of aging, such as fine lines, dark spots, and sagging. Embody's retinol gummy has also the goal to reduce the overall frequency of adult acne and an improvement of overall skin health by promoting hydrated, brightened skin. The study aims to collect self-reported outcomes and photographic images to understand the assessment of the efficacy of treatment from the participant's perspective, and if participants see an improvement in their fine lines, wrinkles, dark spots, and sagging.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18-45 years old
* Must be in good general health
* May experiences adult acne and/or early-stage wrinkles that are not treated by topical or oral prescription drugs/medication
* Must maintain a basic skincare routine
* Must discontinue the use of other dietary supplements
* Must be willing to comply with the requirements of the protocol
* Is able to communicate in English
* Is willing to skip their normal skincare routine
* Must provide written informed consent form (ICF)
* Is willing and able to share feedback and take skin pictures via the used technology portal

Exclusion Criteria:

* Unwilling to provide consent
* Unwilling to skip their normal skincare routine
* Unwilling to follow the routine of the protocol
* Use of other oral retinoids
* Use of prescription medication relevant to the skin
* Undergoing any cosmetic procedures during the study including Botox, laser or chemical treatments
* Deep-set of wrinkles
* History of the following medical conditions or diseases:
* Kidney disease
* Liver disease
* Alcohol abuse
* Use of prescription drug (topical or oral) that is targeted at any sort of skin condition (for example retinoids)
* Any known allergies/sensitivities to nuts

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Skin aging [Time frame: Baseline to 8 weeks] | 8 week intervention period
  Patient reported outcome measures (Scale 0-5 with higher scores representing a better outcome) to assess the reduction of early signs of aging such as fine lines, dark spots, and sagging
Adult acne [Time frame: Baseline to 8 weeks] | 8 week intervention period
  Reduction the overall frequency and intensity of adult acne (Scale 0-5 with higher scores representing a reduction in the appearance of adult acne)

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No